CLINICAL TRIAL: NCT02155101
Title: Monotherapy in Africa: Evaluation of New Therapy
Brief Title: Efficacy and Safety Study of Darunavir for the Treatment of HIV/AIDS
Acronym: MANET
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Liverpool (Other)
Collaborators: Janssen Pharmaceutica (Industry); Chantal Biya International Reference Centre for Research on Prevention and Management of HIV/AIDS (Other Government); Yaounde Central Hospital (Other Government)
Responsible Party: Principal Investigator, Anna Maria Geretti, Principal Investigator, University of Liverpool
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ChantalIRCB
Record Dates: First submitted 2014-06-02; First posted 2014-06-04 (Estimated); Results first posted 2019-09-04 (Actual); Last update posted 2019-09-04 (Actual); Status verified 2019-08

CONDITIONS: HIV/AIDS
Keywords: Efficacy; Safety; Darunavir; HIV-1 RNA level; Cameroon
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Darunavir; Lopinavir; Ritonavir; atazanavir, ritonavir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ART with 2 NRTIs plus LPV/r (or ATV/r) (Active Comparator): 2 nucleos(t)ide reverse transcriptase inhibitors (NRTIs) plus either lopinavir/ritonavir (LPV/r) or atazanavir/ritonavir (ATV/r).
  Interventions: Drug: ART with 2 NRTIs plus LPV/r (or ATV/r)
- Darunavir (Experimental): Dosage form: Darunavir (PREZISTA) is a film coated, oval shaped, light orange 19.1mm tablet, debossed with "400 mg" on one side and TMC on the other side.
  Interventions: Drug: Darunavir

INTERVENTIONS:
Drug: Darunavir — Darunavir (PREZISTA) is a film coated, oval shaped, light orange 19.1mm tablet, debossed with 400 mg on one side and TMC on the other side.
  Other Names: PREZISTA
  Arms: Darunavir
Drug: ART with 2 NRTIs plus LPV/r (or ATV/r) — Patients on second line antiretroviral therapy take 2 NRTIs and either protease inhibitor lopinavir/ritonavir or atazanavir/ritonavir.
  Other Names: NRTI, lopinavir/ritonavir (LPV/r), atazanavir/ritonavir (ATV/r)
  Arms: ART with 2 NRTIs plus LPV/r (or ATV/r)

SUMMARY:
The aim of this pilot study is to assess the feasibility, efficacy and safety of Darunavir/ritonavir 800/100 mg once daily (DRV/r) monotherapy as a switch-maintenance strategy for patients receiving second-line ART at Yaoundé Central Hospital in Cameroon. HIV-infected adults receiving second-line antiretroviral therapy (ART) for ≥3 months with 2 nucleos(t)ide reverse transcriptase inhibitors (NRTIs) plus either lopinavir/ritonavir (LPV/r) or atazanavir/ritonavir (ATV/r) will undergo plasma HIV-1 RNA ("viral") load testing. Those with a viral load below 50 copies/ml (<50 cps/ml) will undergo a repeat test ideally 4-6 weeks later (allowed up to 12 weeks); if the viral load is confirmed as <50 cps/ml the patient will be invited to join the randomised phase of the study. Patients (n=150) will be randomised 1:2 to either continue the current triple ART regimen (n=50) or switch to DRV/r monotherapy (n=100). The primary end-point will be viral load suppression <400 cps/ml at week 24; secondary end-points will be viral load suppression <50 cps/ml at week 12 and week 24, safety, tolerability, and emergence of protease inhibitor (PI) drug-resistance. Patients will continue observational follow-up depending on the treatment arm they are randomized to. After week 48, patients will return to local standard of care. Pharmacokinetics (PK) and pharmacogenomics sub-study to correlate plasma concentrations of DRV to outcomes, HIV-1 drug resistance testing sub study to detect mutants archived at the time of first-line ART failure and measuring HIV DNA load will be performed, as well as a cost-effectiveness analysis will test the hypothesis that savings can be achieved by switching to DRV/r monotherapy without affecting quality of care. The primary virological objective is to evaluate efficacy in terms of the percentage of subjects who have plasma HIV-1 RNA levels <400 cps/ml after 24 weeks of follow-up following a switch to DRV/r monotherapy versus continuing triple therapy containing 2 NRTIs + LPV/r (or ATV/r) (FDA Snapshot method).

Study hypothesis:

we propose that maintenance therapy with DRV/r monotherapy is a feasible, effective and safe treatment option for patients receiving second-line ART in Yaoundé.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with documented HIV-1 infection.
2. Male or female aged > 21 years old.
3. Subjects receiving ART with 2 NRTIs + LPV/r (or ATV/r) for at least 3 months at the time of Screening 1.
4. Nadir T lymphocyte cluster of differentiation 4 (CD4) >100 cells/mm3
5. Plasma HIV-1 RNA <50 copies/ml at Screening 1 confirmed ideally 4-6 weeks later at Screening 2 (two results must be documented; a first result obtained up to 12 weeks earlier will be accepted).
6. Subjects can comply with the protocol requirements. In particular, subjects should be willing to be followed up at least until week 24 (discontinuation prior to week 24) and for the DRV/r arm up to week 48 (discontinuation after week 24) even if they discontinue randomized treatment.
7. Subjects who have voluntarily signed and dated the consent form.

Exclusion Criteria:

1. Clinical or laboratory evidence of significantly decreased hepatic function or decompensation, irrespective of liver enzyme levels (liver insufficiency).
2. Co-infection with hepatitis B (HBsAg positive).
3. Grade 3 or 4 laboratory abnormality as defined by AIDS, including haemoglobin ≤8mg/dL; platelets ≤50 000/mm3; estimated creatinine clearance ≤60ml/ minute, aspartate aminotransferase; alanine aminotransferase and alkaline phosphatase >3 times the upper limit of normal; and total bilirubin >2.5 times the upper limit of normal; with the following exceptions unless clinical assessment foresees an immediate health risk to the subject:

   * Pre-existing diabetes or asymptomatic glucose grade 3 or 4 elevations.
   * Asymptomatic triglyceride or cholesterol elevations of grade 3 or 4.
4. Presence of any currently active AIDS defining illness (Category C conditions according to the Centers for Disease Control Classification System for HIV Infection 1993) with the following exceptions:

   * Stable cutaneous Kaposi's Sarcoma (i.e., no internal organ involvement other than oral lesions) that is unlikely to require any form of systemic therapy during the study.
   * Wasting syndrome due to HIV infection. Note: An AIDS defining illness that is not clinically stabilized for at least 30 days will be considered as currently active.
5. Pregnant or breastfeeding women.
6. Active substance abuse, including alcohol or recreational drugs.
7. Any clinically significant disease (e.g., tuberculosis, cardiac dysfunction, pancreatitis, acute viral infections) or life threatening disease in the previous 14 days, or findings during screening of medical history or physical examination that, in the investigator's opinion, would compromise the subject's safety or outcome of the study.
8. Any medical or psychiatric condition which, in the opinion of the investigator, could compromise the subject's safety or adherence to the trial protocol.
9. Previously demonstrated clinically allergy or hypersensitivity to any of the excipients of the investigational medication (DRV).

   Note: DRV is a sulfonamide. Subjects who have previously experienced a sulfonamide allergy will be allowed to enter the trial. To date, no potential for cross sensitivity between drugs in the sulfonamide class and DRV has been identified in subjects participating in phase II trials.
10. Participation in any other clinical trials that involve administration of antiretrovirals or other drugs within the last 4 weeks and during the participation in this trial.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2014-05; Primary Completion 2016-06 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anna Maria Geretti, MD, PhD, Principal Investigator — University of Liverpool
Locations (1):
- Yaounde Central Hospital, Yaoundé, Centre Region, Cameroon

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Geretti AM, Abdullahi A, Mafotsing Fopoussi O, Bonnett L, Fokom Defo V, Moudourou S, Fokam J, Kouanfack C, Torimiro J. An apparent paradox: resistance mutations in HIV-1 DNA predict improved virological responses to antiretroviral therapy. J Antimicrob Chemother. 2019 Oct 1;74(10):3011-3015. doi: 10.1093/jac/dkz264. PMID 31299067

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ART With 2 NRTIs Plus LPV/r (or ATV/r) | Darunavir
Started | 39 | 81
Completed | 39 | 80
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ART With 2 NRTIs Plus LPV/r (or ATV/r) | Darunavir | Total
Number analyzed (Participants) | 39 | 81 | 120
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 45 [38 to 51] | 45 [37 to 52] | 45 [38 to 52]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 61 | 91
  Male | 9 | 20 | 29
Region of Enrollment [Number; unit: participants]
  Cameroon | 39 | 81 | 120
Body mass index [Median (Inter-Quartile Range); unit: kg/m^2] | 26.0 [22.5 to 29.2] | 25.4 [21.8 to 28.4] | 25.5 [22.1 to 29.1]
Haemoglobin [Median (Inter-Quartile Range); unit: g/dl] | 12.4 [11.6 to 13.5] | 12.3 [11.6 to 13.2] | 12.3 [11.6 to 13.5]
Estimated glomerular filtration rate >90 [Count of Participants; unit: Participants] | 35 | 67 | 102
Time since HIV diagnosis [Median (Inter-Quartile Range); unit: years] | 8.0 [5.5 to 9.8] | 8.8 [5.9 to 11.1] | 8.5 [5.8 to 10.4]
CD4 cell count [Median (Inter-Quartile Range); unit: cells/mm3] | 536 [394 to 687] | 466 [341 to 615] | 467 [341 to 618]
History of previous AIDS defining diagnosis [Count of Participants; unit: Participants] | 4 | 12 | 16
HIV-1 DNA [Median (Inter-Quartile Range); unit: log10 copies/106 PBMC] | 2.7 [2.2 to 2.9] | 2.9 [2.5 to 3.3] | 2.9 [2.4 to 3.2]
Duration on antiretroviral therapy(ART) [Median (Inter-Quartile Range); unit: years] | 6.9 [4.9 to 9.2] | 7.6 [5.3 to 9.8] | 7.5 [5.3 to 9.4]
Duration on protease inhibitor based ART [Median (Inter-Quartile Range); unit: years] | 3.1 [1.5 to 4.9] | 3.2 [1.3 to 5.8] | 3.1 [1.3 to 5.3]
ART regimen at baseline [Count of Participants; unit: Participants]
  Tenofovir/lamivudine + lopinavir/ritonavir | 37 | 69 | 106
  Abacavir + didanosine + lopinavir/ritonavir | 1 | 5 | 6
  Zidovudine/lamivudine + lopinavir/ritonavir | 1 | 4 | 5
  Tenofovir/lamivudine + atazanavir/ritonavir | 0 | 2 | 2
  Tenofovir + abacavir + lopinavir/ritonavir | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: HIV-1 RNA Viral Load
Description: Percentage of subjects who have plasma HIV-1 RNA levels <400 cps/ml after 24 weeks of follow-up following a switch to DRV/r monotherapy versus continuing triple therapy containing 2 NRTIs + LPV/r (or ATV/r) (FDA Snapshot method). The FDA 'Snapshot' algorithm evaluates HIV RNA response using only the results at the week 24 time-point which also means that rebound at earlier time-points are not classified as treatment failure, unless it lead to discontinuation prior to the week 48.
Time Frame: 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | ART With 2 NRTIs Plus LPV/r (or ATV/r) | Darunavir
Number analyzed (Participants) | 39 | 81
Participants | 37 | 72

2. Secondary Outcome: HIV-1 RNA Viral Load
Description: Percentage of subjects who have plasma HIV-1 RNA levels <50 cps/ml after 12 weeks of follow-up following a switch to DRV/r monotherapy versus continuing triple therapy containing 2 NRTIs + LPV/r (or ATV/r), using the FDA "Time to Loss of Virologic Response" method. The FDA 'Snapshot' algorithm evaluates HIV RNA response using only the results at the week 12 time-point which also means that rebound at earlier time-points are not classified as treatment failure, unless it lead to discontinuation prior to the week 48.
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | ART With 2 NRTIs Plus LPV/r (or ATV/r) | Darunavir
Number analyzed (Participants) | 39 | 81
Participants | 35 | 73

3. Other Pre Specified Outcome: HIV-1 RNA Viral Load
Description: Percentage of subjects who have plasma HIV-1 RNA levels <50 cps/ml after 24 weeks of follow-up following a switch to DRV/r monotherapy versus continuing triple therapy containing 2 NRTIs + LPV/r (or ATV/r), using the FDA "Time to Loss of Virologic Response" method. The FDA 'Snapshot' algorithm evaluates HIV RNA response using only the results at the week 24 time-point which also means that rebound at earlier time-points are not classified as treatment failure, unless it lead to discontinuation prior to the week 48.
Time Frame: 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | ART With 2 NRTIs Plus LPV/r (or ATV/r) | Darunavir
Number analyzed (Participants) | 39 | 81
Participants | 36 | 62

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over the 48 week study period
Arm/Group | ART With 2 NRTIs Plus LPV/r (or ATV/r) | Darunavir
All-Cause Mortality (participants affected / at risk) | 0/39 | 1/81
Serious Adverse Events (participants affected / at risk) | 0/39 | 3/81
Other Adverse Events (participants affected / at risk) | 2/39 | 3/81
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ART With 2 NRTIs Plus LPV/r (or ATV/r) (N=39) | Darunavir (N=81)
Car accident, hospitalisation, resolved; (Social circumstances) | NA | 1 (1)
acute anxiety, hospitalisation, resolved (General disorders) | NA | 1 (1)
malaria, progressive anaemia, hospitalisation, transfusion reaction, death (Infections and infestations) | NA | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ART With 2 NRTIs Plus LPV/r (or ATV/r) (N=39) | Darunavir (N=81)
Acute hepatitis B (Infections and infestations) | 0 (0) | 1 (1)
Acute febrile illness (General disorders) | 1 (1) | 0 (0)
Hypertension (General disorders) | 1 (1) | 1 (1)
Pulmonary TB (Infections and infestations) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less